CLINICAL TRIAL: NCT00297765
Title: OPTIMA (Optimizing Prograf® Therapy in Renal Transplant Patients)
Brief Title: Optimizing Prograf® Therapy in Renal Transplant Patients
Acronym: OPTIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-02-002
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2007-12

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Therapeutics; Treatment Outcome; Safety
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tacrolimus, Prograf®

SUMMARY:
A study to determine the optimal dose and blood level of Prograf® in long-term maintenance of kidney transplant patients.

DETAILED DESCRIPTION:
A 3 arm study (2 Active, 1 Active Control) to determine the optimal dose and blood level of Prograf® in long-term maintenance of kidney transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Patient was 18 years of age at the time of transplant.
* Patient is at least 6 months post-transplant.

Exclusion Criteria:

* Patient is the recipient of a solid organ transplant other than the kidney.
* Patient is a known carrier of any of the HIV viruses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2003-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The effect of conversion from cyclosporine to Prograf-based therapy on renal function | 12 months

SECONDARY OUTCOMES:
Assessment of renal function, Cystatin C, TGF-beta, biopsy proven rejection, and patient and graft survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John Holman, MD, Study Director — Astellas Pharma US, Inc.
Locations (37):
- United States (37):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Portland, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Livingston, New Jersey
  - West Orange, New Jersey
  - Buffalo, New York
  - Long Island City, New York
  - Mineola, New York
  - New York, New York
  - Greenville, North Carolina
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington